CLINICAL TRIAL: NCT04748016
Title: Sterilised 3D-PRINTed Bone Models in Addition to Conventional CT Imaging for Operative Visualisation in Complex Intra-articular Fracture Repair - A Multi-centre, Double-blind Randomised Controlled Trial
Brief Title: 3D-printed Bone Models in Addition to CT Imaging for Intra-articular Fracture Repair
Acronym: SPRINT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Christian Xinshuo Fang, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 18-480
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Distal Humerus Fracture; Distal Femur Fracture; Distal Tibia Fracture; Proximal Humeral Fracture
Keywords: 3D Printing; Intra-articular Fracture; Patient-specific instrumentation
MeSH Terms: conditions — Humeral Fractures, Distal; Femoral Fractures, Distal; Shoulder Fractures; Intra-Articular Fractures | interventions — Postmortem Imaging

STUDY DESIGN:
Intervention Model Description: Double-blind randomised control trial with 40 patients in two interventional arm
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are randomly assigned to either one of the interventional arm and will not be informed of the randomisation result.
  A blinded reviewer will assess the postoperative radiographs and surgical quality.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-printed models plus CT imaging (Experimental): Fracture repair surgery using sterilized 3DP models, CT-MPR and CT-3DR for planning and intraoperative visualization
  Interventions: Other: 3D printed (3DP) bone models + CT imaging
- CT imaging alone (Active Comparator): Fracture repair surgery using CT-MPR and CT-3DR for planning and intraoperative visualization
  Interventions: Other: CT imaging

INTERVENTIONS:
Other: 3D printed (3DP) bone models + CT imaging — In addition to CT-MPR and CT-3DR, 3DP models will be used for surgical planning and intraoperative visualization.
  Arms: 3D-printed models plus CT imaging
Other: CT imaging — CT-MPR and CT-3DR used for surgical planning and intraoperative visualization.
  Arms: CT imaging alone

SUMMARY:
The purpose of this study is to compare the effectiveness of 3D-printed bone models in addition to CT imaging versus CT imaging alone on surgical quality and operation time for patients undergoing surgical repair of intra-articular fractures.

DETAILED DESCRIPTION:
Surgical fixation of intra-articular fractures is a technically demanding task that poses significant challenges to orthopaedic surgeons. Articular fragments may be comminuted, depressed, or impacted, and neighbouring soft tissue is often heavily compromised. Furthermore, aggressive surgical dissection is typically necessary to achieve adequate visualisation, and anatomical reduction often devitalises bone fragments and invites deep infection. The management of intra-articular fractures requires a well-designed preoperative plan and a skilfully executed surgical tactic to guarantee the best possible outcome. Multiplanar reformation (CT-MPR) and three-dimensional reconstruction (CT-3DR) are imaging techniques that have enhanced intraoperative visualisation, however, accurate analysis of complex fractures remains challenging.

3D printing is a rapidly developing, low-cost technology that is already being applied across numerous contexts in orthopaedics and traumatology. 3D printed bone models can be produced from digitised CT data in a matter of hours, providing a dimensionally accurate representation of the patient's skeleton which approximates real-life visual and tactile experiences. When used in preoperative planning, these models have shown to improve surgeon communication and shorten surgical duration. Despite positive early results, few clinical studies have studied the effect of 3D bone model use on surgical outcome. The purpose of this randomised controlled trial is to compare the effectiveness of intraoperatively utilised 3D bone models in addition to conventional CT imaging on reduction quality and surgical duration versus CT imaging alone for patients undergoing surgical fixation of complex intraarticular fractures.

Patients providing informed consent will be screened for eligibility. All eligible patients will be randomly assigned in a double-blind manner (participant and outcome assessor) to receive surgical fracture fixation with or without the addition of sterilised 3D-printed bone models to standard CT imaging for intraoperative visualisation.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or older
2. with intra-articular fracture of the proximal or distal humerus, proximal ulna, proximal radius, distal femur, or proximal or distal tibia (pilon fracture)
3. requiring anticipated surgical repair of fracture
4. with pre-operative CT scan already available as part of routine assessment

Exclusion Criteria:

1. pathological fracture
2. multiple fractures requiring simultaneous or staged operations
3. fractures around the hip, pelvis and acetabulum, and any other fracture types not specified in the inclusion criteria
4. requiring surgery within 24 hours of admission
5. unable or unwilling to give consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of articular surface reduction grading assessed by three-point scale | Immediately post-operation
  The quality of articular surface reduction will be rated by two surgeons blinded to intervention allotment assessing post-operative and intraoperative fluoroscopic images. The Kappa value will be recorded for inter-observer agreement between two observers (1. Perfect reduction, 2. Observable imperfections 1-2mm, 3. Significant imperfections >2mm)
Skin to skin duration of surgery (minutes) | Immediately post-operation
  The skin to skin duration of the surgery will be recorded.

SECONDARY OUTCOMES:
Total fluoroscopy time (seconds) | Immediately post-operation
  The total intraoperative fluoroscopy time will be recorded in seconds.
Intraoperative blood loss (mL) | Immediately post-operation
  The patient's blood loss during the surgery will be recorded.
Total length of skin incision (mm) | Immediately post-operation
  The total length on the incision will be measured post operation.
Total tourniquet time (minutes) | Immediately post-operation
  Total time the tourniquet was applied will be recorded.
Incidence of surgical complications | 3 months post-operation
  Incidence of infection, neurological deficit, wound breakdown, loss of fixation, revision surgery will be recorded at follow up.
Quality of articular surface reduction grading assessed by three-point scale | 3 months post operation
  The quality of articular surface reduction will be rated by two surgeons blinded to intervention allotment assessing post-operative and intraoperative fluoroscopic images. The Kappa value will be recorded for inter-observer agreement between two observers (1. Perfect reduction, 2. Observable imperfections 1-2mm, 3. Significant imperfections >2mm)
Health-related quality of life measured by SF-12 Chinese (HK) version | 3 months post-operation
  12-item Short Form Health Survey (SF-12), a patient-reported outcome measure of HRQOL comprised of a mental component (MCS) and physical component (PCS), each with a final score ranging from 0 (worst outcome) to 100 (best outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Christian Fang, Principal Investigator — Dept of Orthopaedics and Traumatology, Queen Mary Hospital
Locations (1):
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Anonymized dataset to be included as supplementary data in final publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 1 year of study completion
Access Criteria: Additional information available upon reasonable request of principal investigator

REFERENCES:
- [Background] Jupiter JB, Fernandez DL, Toh CL, Fellman T, Ring D. Operative treatment of volar intra-articular fractures of the distal end of the radius. J Bone Joint Surg Am. 1996 Dec;78(12):1817-28. doi: 10.2106/00004623-199612000-00004. PMID 8986658
- [Background] Kang HW, Lee SJ, Ko IK, Kengla C, Yoo JJ, Atala A. A 3D bioprinting system to produce human-scale tissue constructs with structural integrity. Nat Biotechnol. 2016 Mar;34(3):312-9. doi: 10.1038/nbt.3413. Epub 2016 Feb 15. PMID 26878319
- [Background] You W, Liu LJ, Chen HX, Xiong JY, Wang DM, Huang JH, Ding JL, Wang DP. Application of 3D printing technology on the treatment of complex proximal humeral fractures (Neer3-part and 4-part) in old people. Orthop Traumatol Surg Res. 2016 Nov;102(7):897-903. doi: 10.1016/j.otsr.2016.06.009. Epub 2016 Aug 9. PMID 27521179
- [Background] Yang L, Shang XW, Fan JN, He ZX, Wang JJ, Liu M, Zhuang Y, Ye C. Application of 3D Printing in the Surgical Planning of Trimalleolar Fracture and Doctor-Patient Communication. Biomed Res Int. 2016;2016:2482086. doi: 10.1155/2016/2482086. Epub 2016 Jul 3. PMID 27446944
- [Background] Kacl GM, Zanetti M, Amgwerd M, Trentz O, Seifert B, Stucki H, Hodler J. Rapid prototyping (stereolithography) in the management of intra-articular calcaneal fractures. Eur Radiol. 1997;7(2):187-91. doi: 10.1007/s003300050132. PMID 9038112
- [Background] Yan CH, Chiu KY, Ng FY, Chan PK, Fang CX. Comparison between patient-specific instruments and conventional instruments and computer navigation in total knee arthroplasty: a randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2015 Dec;23(12):3637-45. doi: 10.1007/s00167-014-3264-2. Epub 2014 Sep 13. PMID 25217311
- [Background] Yang J, Cai H, Lv J, Zhang K, Leng H, Sun C, Wang Z, Liu Z. In vivo study of a self-stabilizing artificial vertebral body fabricated by electron beam melting. Spine (Phila Pa 1976). 2014 Apr 15;39(8):E486-92. doi: 10.1097/BRS.0000000000000211. PMID 24430723
- [Background] Peltola SM, Melchels FP, Grijpma DW, Kellomaki M. A review of rapid prototyping techniques for tissue engineering purposes. Ann Med. 2008;40(4):268-80. doi: 10.1080/07853890701881788. PMID 18428020
- [Background] Brown GA, Firoozbakhsh K, DeCoster TA, Reyna JR Jr, Moneim M. Rapid prototyping: the future of trauma surgery? J Bone Joint Surg Am. 2003;85-A Suppl 4:49-55. No abstract available. PMID 14652393
- [Background] Hurson C, Tansey A, O'Donnchadha B, Nicholson P, Rice J, McElwain J. Rapid prototyping in the assessment, classification and preoperative planning of acetabular fractures. Injury. 2007 Oct;38(10):1158-62. doi: 10.1016/j.injury.2007.05.020. Epub 2007 Sep 19. PMID 17884058
- [Background] Bizzotto N, Tami I, Tami A, Spiegel A, Romani D, Corain M, Adani R, Magnan B. 3D Printed models of distal radius fractures. Injury. 2016 Apr;47(4):976-8. doi: 10.1016/j.injury.2016.01.013. Epub 2016 Feb 6. No abstract available. PMID 26876530
- [Background] Li Z, Li Z, Xu R, Li M, Li J, Liu Y, Sui D, Zhang W, Chen Z. Three-dimensional printing models improve understanding of spinal fracture--A randomized controlled study in China. Sci Rep. 2015 Jun 23;5:11570. doi: 10.1038/srep11570. PMID 26099838
- [Background] Fang C, Fang B, Wong TM, Lau TW, Pun T, Leung F. Fixing a fractured arthrodesed hip with rapid prototype templating and minimal invasive plate osteosynthesis. Trauma Case Rep. 2015 Nov 14;1(9-12):79-83. doi: 10.1016/j.tcr.2015.10.005. eCollection 2015 Dec. PMID 30101181
- [Background] Wong TM, Jin J, Lau TW, Fang C, Yan CH, Yeung K, To M, Leung F. The use of three-dimensional printing technology in orthopaedic surgery. J Orthop Surg (Hong Kong). 2017 Jan;25(1):2309499016684077. doi: 10.1177/2309499016684077. PMID 28142354
- [Background] Fedorov A, Beichel R, Kalpathy-Cramer J, Finet J, Fillion-Robin JC, Pujol S, Bauer C, Jennings D, Fennessy F, Sonka M, Buatti J, Aylward S, Miller JV, Pieper S, Kikinis R. 3D Slicer as an image computing platform for the Quantitative Imaging Network. Magn Reson Imaging. 2012 Nov;30(9):1323-41. doi: 10.1016/j.mri.2012.05.001. Epub 2012 Jul 6. PMID 22770690
- [Background] Suresh K. An overview of randomization techniques: An unbiased assessment of outcome in clinical research. J Hum Reprod Sci. 2011 Jan;4(1):8-11. doi: 10.4103/0974-1208.82352. PMID 21772732
- [Background] Rennie D. CONSORT revised--improving the reporting of randomized trials. JAMA. 2001 Apr 18;285(15):2006-7. doi: 10.1001/jama.285.15.2006. No abstract available. PMID 11308440
- [Background] Zarin DA, Tse T, Williams RJ, Califf RM, Ide NC. The ClinicalTrials.gov results database--update and key issues. N Engl J Med. 2011 Mar 3;364(9):852-60. doi: 10.1056/NEJMsa1012065. PMID 21366476